CLINICAL TRIAL: NCT05962970
Title: Continuous Adductor Canal Block in Fast Track Total Knee Arthroplasty
Acronym: CACB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Principal Investigator, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-0041-A
Record Dates: First submitted 2023-06-08; First posted 2023-07-27 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Total Knee Arthroplasty
Keywords: Orthopaedic; Postoperative Pain Management; total knee arthroplasty; Continuous adductor canal block; Fast-track
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CACB (Active Comparator): continuous adductor canal block
  Interventions: Drug: continuous adductor canal block (CACB) ropivacaine
- Control group (Placebo Comparator): sham continuous adductor canal block - ShACB
  Interventions: Drug: sham continuous adductor canal block - ShACB NaCl

INTERVENTIONS:
Drug: continuous adductor canal block (CACB) ropivacaine — The CACB group will receive an infusion of 0.2% ropivacaine 5mL/h
  Arms: CACB
Drug: sham continuous adductor canal block - ShACB NaCl — sham continuous adductor canal block - ShACB and ShACB group will receive an infusion of NaCl 0.9% 5mL/h.
  Arms: Control group

SUMMARY:
Total knee arthroplasty (TKA) is a frequent performed surgery. Many institutions are implementing fast track programs for this surgery and adequate pain management is an important feature. Analgesic duration of single shot nerve blocks is limited to no more than 24h. Conversely, the use of continuous nerve block (CNB) through a perineural catheter and infusion of local anesthetic may increase duration of analgesia and provide better outcomes. The purpose of this study is to evaluate effectiveness and safety of using CNB in patients undergoing ambulatory TKA, and its effects on patients' quality of recovery. Investigators hypothesize that continuous adductor canal block would lead to decrease in opioid consumption in patients undergoing fast track TKA.

Significance There are no published prospective randomized controlled trials to assess patient's reported quality of recovery after receiving CACB in same day primary knee arthroplasties. As this is a frequent type of surgery and has the prediction to increase its incidence for the next years, there is significant importance in investigations about interventions which may improve its recovery in a fast track regime. A postoperative analgesic technique that offers better pain control, has less adverse effects, reduces the opioid analgesia requirement and is safe to be used in a fast track setting may have additional impact on decreasing health care cost and may lead to an enhanced recovery and better quality of life.

Objectives To evaluate effectiveness and safety of using CACB in patients undergoing ambulatory TKA, in comparison to SACB. Primary objective is opioid consumption (in oral morphine equivalent doses) Secondary objectives are to evaluate postoperative QoR-15 scores (10), pain scores, opioid-induced adverse effects (measured via validated opioid symptom distress scale), postoperative functional status, complications relating to the perineural catheter and readmissions.

DETAILED DESCRIPTION:
Objectives The aim of this study is to examine the effect of CACB on decreasing opioid consumption, increasing the Quality of Recovery (measured via QoR-15) total score and decreasing opioid-related side effects. Investigators will also assess the rate of readmissions in primary knee arthroplasty patients.

Rationale

Pain management in knee arthroplasty patients poses unique challenges for the anesthesiologist, especially in the immediate post-operative period. Early postoperative analgesia is limited to a unimodality of intravenous opioids. Recently, adductor canal blocks have started to replace femoral blocks, as this technique can provide similar analgesic results while avoiding the quadriceps muscle weakness associated with femoral nerve blocks. The use of a continuous adductor canal catheter in the post-discharge phase shows promising as the next step in knee arthroplasty pain management allowing for shorter lengths of stay or even same day discharge (3).

Significance and Innovation

Total knee arthroplasty (TKA) is the second most common inpatient surgery in the U.S. and Canada, and is associated with severe postoperative pain, limiting early ambulation and optimal functional recovery. Perioperative opioid use has been linked with many adverse outcomes including opioid dependence. This study aims to demonstrate the utility of CACB as an adjunct strategy to reduce opioid consumption and improve quality of recovery in primary knee arthroplasty patients. The innovation in this approach lies not only in less opioid consumption and opioid induced side effects but also in reducing the burden of postoperative pain, leading to an enhanced recovery and better quality of life. Establishing the safeness of this method in an outpatient setting may have the additional impact of decreasing health care costs and may lead to reduce opioid prescriptions on discharge from the hospital.

This will be the first study assessing patient's reported quality of recovery after receiving CACB for primary knee arthroplasties. Investigators expect that that the use of CACB will improve patients' quality of recovery, alleviate pain and also reduce opioid consumption and side effects.

Methodology

This will be a prospective, randomized double blind placebo controlled clinical trial. There will be two arms of treatment: intervention and control group. Preoperatively patients will be allocated at random to receive either Continuous adductor canal block (CACB) (intervention group) or sham continuous adductor canal block (ShACB) (control group).

Work Plan

This prospective trial would include unilateral primary TKA done under Fastrack protocol. The subjects will have their surgeries booked in advance and they will be submitted to the pre anesthesia consult at the Pre-Admission Unit a few days before the surgery. The study proposal will be explained to the patients at time of preadmission consult. They will receive a booklet with information about the study and the Consent Form that they will bring home with them. Patients will be randomized to one of the two groups using a computer-generated random numbers table. The elastomeric pumps to be used connected to the catheter will be previously prepared by hospital pharmacy, accordingly to the randomization made and the subject study number, with no identification of the content (NaCl 0.9% or Ropivacaine 0.2%). All patients will receive the same perioperative management. The only difference will be the postoperative continuous perineural infusion: the CACB group will receive an infusion of 0.2% ropivacaine 5mL/h and ShACB group will receive an infusion of NaCl 0.9% 5mL/h. Patients will initially be brought to a dedicated block room where a safety checklist will be performed by the block room team before performing the block. Standard Canadian Anesthesia Society monitoring will be provided. After surgery, the patient will be taken to the Post Anesthesia Care Unit. At this moment, an Arrow® (StimuCath® Continuous Peripheral Nerve Block Catheter) continuous adductor canal block catheter will be inserted using a Sonosite Edge II ultrasound machine. The patient may be discharged home after achieving the discharge criteria, keeping the peripheral nerve catheter with the same infusion rate for the planned time. The adductor canal catheter will infuse for 48 hours. Prior to going home, patients will receive education and written information (educational pamphlet) regarding monitoring for local anesthetic systemic toxicity symptoms, possible CABC associated complications including potential transient muscle weakness, and instructions on patient removal of the catheter after 48 hours. The study coordinator will collect the data once a day at 24, 48, 72 hrs, seven, 30 and 90 days postoperatively. Data collection will require at maximum 15 minutes.

Sample Size Sample size justification was based on the primary outcome, and the primary objective. The sample size was calculated based on previous study (12) that showed a 48-hour opioid consumption of 30mg (+/- 15 mg) morphine equivalents in knee replacement surgeries at our institute. Investigators anticipate a 50% decrease of opioid use in the intervention group with an alpha of 0.05, power of 80%, and an enrolment ratio of 1:1 (between the 2 groups). This will require 16 subjects in each group for a total of 32 patients. To compensate for 15 to 20% anticipated dropouts from the study, investigators plan for an inclusion of 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TKA in the fast track setting.
* Patients older than 21 years of age, with American Society of Anesthesiologists (ASA)
* Physical status I-III
* No alcohol or drug dependency
* Sufficient understand and co-operation about the perineural catheter.

Exclusion Criteria:

* Perioperative complication or discharge delay leading to hospital admission.
* Chronic opioid use of morphine 30mg equivalent per day for last 2 consecutive weeks.
* Allergy to the study medications;
* Coagulopathy and platelet count < 105/μL;
* Patients with contraindications to the insertion of an epidural or adductor canal catheter (severe anatomic abnormalities or history of previous surgery at the site of catheter placement).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-08-03 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively
  opioid consumption. Total opioid consumption changes will be assessed at 24, 48, 72 hours, seven, 30 and 90 days postoperatively.

SECONDARY OUTCOMES:
Quality of Recovery | At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively
  Quality of Recovery (via QoR-15) total score. Changes will be assessed via QoR-15 (Quality of Recovery). (From score 0 to 10, higher scores mean a better outcome .(At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively)
Intensity of postoperative pain | At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively
  The intensity of postoperative pain. Changes will be assessed by Visual Analog Scale (VAS) at rest and movement once a day using a categorical pain scoring system. (From score 0 to 10, higher scores mean a worse outcome) (At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively)
Opioid related side effects | At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively
  Opioid related side effects. Changes will be assessed using Opioid-related symptom Distress Scale (ORSDS). (At baseline, 24, 48, 72 hours, seven, 30 and 90 days postoperatively)

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — Associate Professor
Locations (1):
- Mount Sinai Hospital, Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, Carr A, Beard D. Knee replacement. Lancet. 2018 Nov 3;392(10158):1672-1682. doi: 10.1016/S0140-6736(18)32344-4. PMID 30496082
- [Background] Cullom C, Weed JT. Anesthetic and Analgesic Management for Outpatient Knee Arthroplasty. Curr Pain Headache Rep. 2017 May;21(5):23. doi: 10.1007/s11916-017-0623-y. PMID 28283810
- [Background] Wang J, Vahid S, Eberg M, Milroy S, Milkovich J, Wright FC, Hunter A, Kalladeen R, Zanchetta C, Wijeysundera HC, Irish J. Clearing the surgical backlog caused by COVID-19 in Ontario: a time series modelling study. CMAJ. 2020 Nov 2;192(44):E1347-E1356. doi: 10.1503/cmaj.201521. Epub 2020 Sep 1. PMID 32873541
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648
- [Background] Leung P, Dickerson DM, Denduluri SK, Mohammed MK, Lu M, Anitescu M, Luu HH. Postoperative continuous adductor canal block for total knee arthroplasty improves pain and functional recovery: A randomized controlled clinical trial. J Clin Anesth. 2018 Sep;49:46-52. doi: 10.1016/j.jclinane.2018.06.004. Epub 2018 Jun 8. PMID 29890381
- [Background] Yu R, Wang H, Zhuo Y, Liu D, Wu C, Zhang Y. Continuous adductor canal block provides better performance after total knee arthroplasty compared with the single-shot adductor canal block?: An updated meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Oct 23;99(43):e22762. doi: 10.1097/MD.0000000000022762. PMID 33120783
- [Background] Hanson NA, Lee PH, Yuan SC, Choi DS, Allen CJ, Auyong DB. Continuous ambulatory adductor canal catheters for patients undergoing knee arthroplasty surgery. J Clin Anesth. 2016 Dec;35:190-194. doi: 10.1016/j.jclinane.2016.07.022. Epub 2016 Aug 30. PMID 27871518
- [Background] Myles PS. More than just morbidity and mortality - quality of recovery and long-term functional recovery after surgery. Anaesthesia. 2020 Jan;75 Suppl 1:e143-e150. doi: 10.1111/anae.14786. PMID 31903564
- [Background] Sun C, Zhang X, Song F, Zhao Z, Du R, Wu S, Ma Q, Cai X. Is continuous catheter adductor canal block better than single-shot canal adductor canal block in primary total knee arthroplasty?: A GRADE analysis of the evidence through a systematic review and meta-analysis. Medicine (Baltimore). 2020 May;99(20):e20320. doi: 10.1097/MD.0000000000020320. PMID 32443383
- [Background] Khan MI, Khandadashpoor S, Rai Y, Vertolli G, Backstein D, Siddiqui N. Comparing Analgesia on an As-Needed Basis to Traditional Intravenous Patient-Controlled Analgesia Within Fast-Track Orthopedic Procedures: A Randomized Controlled Trial. Pain Manag Nurs. 2022 Dec;23(6):832-837. doi: 10.1016/j.pmn.2022.04.003. Epub 2022 May 20. PMID 35599141